CLINICAL TRIAL: NCT02835794
Title: A Phase I/II Clinical Trial of Omacetaxine, Azacitidine, and G-CSF for Relapsed and/or Refractory Myelodysplastic Syndromes
Brief Title: A Clinical Trial of Omacetaxine, Azacitidine, and Growth-Colony Stimulating Factor (G-CSF) for Myelodysplastic Syndromes (MDS)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding to support clinical trial
Sponsor: University of Florida (Other)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601194; UF-MDS-OAG-101 (Other: UF)
Record Dates: First submitted 2016-06-30; First posted 2016-07-18 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Homoharringtonine; Azacitidine; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Omacetaxine - escalating doses subcutaneous twice daily on Days 1-5 and 8-12 Azacitidine 50 mg/m2 subcutaneous/intravenous daily on Days 8-12 G-CSF 5mcg/kg subcutaneous daily on Days 15-19 and 22-26
  Interventions: Drug: Omacetaxine; Drug: Azacitidine; Drug: G-CSF

INTERVENTIONS:
Drug: Omacetaxine — Comparison of different doses of omacetaxine in combination with azacitidine and G-CSF
  Other Names: Synribo
Drug: Azacitidine — Comparison of different doses of omacetaxine in combination with azacitidine and G-CSF
  Other Names: Vidaza
Drug: G-CSF — Comparison of different doses of omacetaxine in combination with azacitidine and G-CSF
  Other Names: Neupogen

SUMMARY:
The purpose of this study is to determine the safety and establish the maximum tolerated dose (MTD) of omacetaxine in combination with azacitidine and G-CSF in patients with relapsed and/or refractory MDS.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* Informed consent;
* Low- and intermediate-risk MDS that has failed to achieve any hematologic improvement after at least 4 cycles of induction therapy or has relapsed after any duration of any hematologic response. Prior therapy with azanucleosides (i.e., azacitidine, decitabine), biologic therapies (i.e., lenalidomide, rigosertib) and hematopoietic cell transplant are permissible;
* Performance status must be Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2;
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) may participate, provided they meet the following conditions:

  * Must agree to use physician-approved contraceptive methods throughout the study and for three months following the last dose of omacetaxine and
  * Must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this trial;
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods throughout the study and should avoid conceiving a child for 6 months following the last dose of omacetaxine.

Exclusion Criteria:

* Subjects who are eligible for hematopoietic stem cell transplant;
* History of atrial fibrillation related to azanucleoside therapy in the past;
* Active, uncontrolled, clinically significant infection;
* Pregnant and nursing patients are excluded because the effects of omacetaxine on a fetus or nursing child are unknown;
* Treatment with any anticancer therapy (standard or investigational) within the previous 14 days prior to the first dose of study drug or less than full recovery from the clinically significant toxic effects of that treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of omacetaxine in combination with azacitidine and G-CSF in patients with relapsed and/or refractory low- and intermediate-risk MDS. | 28 days

SECONDARY OUTCOMES:
Number of participants with Hematologic Improvement (HI) as measured by hemoglobin, platelet count and neutrophil count. | 12 months
Number of participants with disease response as defined by International Working Group (IWG) 2006 criteria. | 12 months
Number of participants who achieve complete remission and how long the response lasts | 24 months
Length of time of survival for participants | 24 months
Incidences of Grade 3/4 adverse events directly related to the drug combination | 24 months

OTHER OUTCOMES:
Number of participants who demonstrate changes in chromosome karyotype and genetic mutations | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maxim N. Norkin, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Shands Cancer Hospital, Gainesville, Florida, United States